CLINICAL TRIAL: NCT07140861
Title: Effect of Core Stability Exercises on Medial Longitudinal Arch Height and Balance in Individuals With Bilateral Flexible Flat Foot
Brief Title: Effect of Core Stability Exercises in Individuals With Bilateral Flexible Flat Foot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Rafat, Assistant professor of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Physical Therapy 52043
Record Dates: First submitted 2025-07-23; First posted 2025-08-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Flat Feet
Keywords: core stability exercises; medial longitudinal arch height; balance; bilateral flexible flat foot
MeSH Terms: conditions — Flatfoot | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group will receive conventional treatment
  Interventions: Other: Conventional
- Study group (Experimental): Study group: will receive core training protocol and conventional therapy.
  Interventions: Other: Conventional; Other: Experimental

INTERVENTIONS:
Other: Conventional — patients will receive conventional therapy that include
  1. Short foot exercises
  2. Towel-curl exercise
  3. Heel raise exercise
  4. Calf stretch
Other: Experimental — Core stability exercises:
  The training programs will last 6 weeks and comprise 3 training sessions per week. Each training session lasted 30 min, starting with a brief, standardized warm-up program mainly consisting of low-intensity core strength exercises to prepare the neuromuscular system for the training loads and ending with a cool-down program (i.e., dynamic stretching). During the main part of training, research group will conduct the "big 3" exercises as described by McGill (Mcgill, 2001). These include the curl-up, side bridge, and quadruped position. In other words, every single training session consisted of frontal, dorsal, and lateral core exercises. Training intensity will be progressed and individually increased over the 6-week training program by modulating lever lengths, movement velocity
  Arms: Study group

SUMMARY:
There is a gap of literature about the role of core stability exercises on management of flexible flatfoot, as a result this study will take a deeper look on the effect of core stability exercises on navicular height, Arch height index, balance and disability function of ankle joint in individuals with bilateral flexible flat foot.

DETAILED DESCRIPTION:
It was proved that Individuals with flexible flat foot have reduced core stability. Thus, core stability must be assessed while treating individuals with flexible flat foot and interventions that address core stability must be included in the treatment of flexible flat foot . It was demonstrated that there was a poorer balance in individual with bilateral flexible flat foot. Therefore, it is recommended to add balance training exercises to traditional physical therapy program in cases of flatfoot patients .

40 Participants of both genders with bilateral flexible flatfoot. will be assigned randomly into 2 equal groups: Group A (control group): will receive conventional therapy. Group B (Experimental group): will receive core training protocol and conventional therapy. Subjects will receive 3 sessions per week for 6 weeks.

Outcome measures:

1. Navicular height: will be evaluated by navicular drop test.
2. Medial longitudinal arch height: will be evaluated by Arch height index (AHI).
3. Balance: will be evaluated by Biodex Balance System.
4. Disability function of ankle joint: will be evaluated by Arabic version of foot function index scale.

ELIGIBILITY:
Inclusion Criteria:

1. 40 Participants of both genders with bilateral flexible flatfoot.
2. Their age ranges from 18 to 39 years.
3. All Participants with a navicular drop (ND) greater than 10 mm.
4. Body mass index from 18.5-25 kg/m2

Exclusion Criteria:

1. Traumatic condition of the lower limbs.
2. History of Fracture of the lower limbs.
3. previous orthopedic disorders or neurologic deficit of the lower limbs.
4. Previous surgery of the lower limbs.
5. Any sensory problems.
6. Leg length discrepancy.
7. Neuromuscular disease like multiple scelerosis.
8. Unilateral flexible flat foot.
9. Rigid flat foot.
10. Any lumbar spine problems

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Navicular height | at enrollment and at the end of 6 weeks of treatment
Balance | at enrollment and at the end of 6 weeks of treatment
  Dynamic balance will be assessed by Biodex system

SECONDARY OUTCOMES:
Medial longitudinal arch height | at enrollment and at the end of 6 weeks of treatment
Function of ankle joint | at enrollment and at the end of 6 weeks of treatment
  Function of ankle joint will be assessed by Arabic version of foot function index scale.

CONTACTS AND LOCATIONS:
Overall Officials: Magda Gaid Professor of physical therapy - Cairo University, Study Director — Department of Basic sciences for physical therapy, Faculty of Physical Therapy , Cairo university, Cairo, Egypt; Ahmed Abdou, Assistant lecturer, Principal Investigator — Department of Basic sciences for physical therapy, Faculty of Physical Therapy , Cairo university, Cairo, Egypt
Locations (2):
- Egypt (2):
  - Physical therapy College - Cairo university, Cairo
  - Physical Therapy faculty, Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: No